CLINICAL TRIAL: NCT06653387
Title: A Multicenter, Single-arm, Pivotal Study to Evaluate Acute Device and Technical Success of the CGuard Prime Carotid Stent System (80cm) When Used in Conjunction With the FDA-cleared ENROUTE Transcarotid Neuroprotection System (NPS) in Patients at High Risk for Adverse Events From Carotid Endarterectomy Undergoing Carotid Artery Stenting Via the Transcarotid Artery Revascularization (TCAR) Approach.
Brief Title: A Single-arm, Pivotal Study to Evaluate Acute Device and Technical Success of the CGuard Prime Carotid Stent System When Used in Conjunction to the ENROUTE Transcarotid Neuroprotection System in Patients Undergoing Carotid Artery Stenting Via the Transcarotid Artery Revascularization Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InspireMD (Industry)
Collaborators: Washington University School of Medicine (Other); TriHealth Inc. (Other); NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGUARDIANS II
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Carotid Artery Diseases
Keywords: Carotid Artery Stenosis; Transcarotid Artery Revascularization; Carotid Artery Angioplasty; Stenting Procedure
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGuard Prime 80cm stent system with ENROUTE NPS (Experimental)
  Interventions: Device: CGuard Prime 80cm stent system

INTERVENTIONS:
Device: CGuard Prime 80cm stent system — This study is single arm looking at the technical success of the CGuard Prime 80cm stent system when used in conjunction with the FDA-cleared ENROUTE NPS during a TCAR procedure.

SUMMARY:
The objective of this study is to evaluate acute device and technical success of the CGuard Prime™ Carotid Stent System (80cm) when used in conjunction with the Enroute NPS during Transcarotid Artery Revascularization procedures in the treatment of carotid artery stenosis in spatients at high risk for adverse events from carotid endarterectomy.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single arm pivotal study. The study shall not be blinded prior to, during or following the procedure. Patients undergoing transcarotid artery revascularization will be screened against the study inclusion/exclusion criteria. If the patient meets study eligibility requirements, they shall be invited to participate, provide informed consent and shall subsequently be assigned a study ID number.

Enrollment will be a minimum of 50 evaluable pivotal patients. A maximum of 20% of patients will be enrolled at any single site. The total enrollment accounts for an estimate that up to 2 patients will exit the study prior to the 30-day primary endpoint assessment.

An additional roll-in cohort of up to 2 patients per primary physician operator at each study site may also be accrued (maximum of 24 roll-in patients total, assuming one primary physician operator per site).

This study does not duplicate any current knowledge existing today on use of the CGuard Prime™ 80 used in conjunction with the ENROUTE NPS in the United States.

ELIGIBILITY:
INCLUSION CRITERIA: Candidates for participation in the study must meet all of the following general inclusion criteria.

* Patient is ≥ 18 years and < 80 years of age.
* Patient is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
* Patient is diagnosed with carotid artery disease treatable with a Carotid Artery Stent via a Transcarotid Artery Revascularization approach and is either symptomatic or asymptomatic, defined as:
* Symptomatic carotid stenosis ≥ 50%. Symptomatic is defined as amaurosis fugax, transient ischemia attack (TIA) or stroke within the last 6 months ipsilateral to the side of the stenosis Or
* Asymptomatic carotid stenosis ≥ 80%
* High Risk condition for CEA: at least one, as shown below:

Comorbid conditions:

* Age ≥ 70 (maximum 80 years)
* CCS angina class 3-4 or unstable angina
* Congestive Heart Failure (CHF) NYHA class III-IV
* Left ventricular ejection fraction (LVEF) ≤ 35%
* MI ≥ 72 hours and < 6 weeks pre-procedure
* Multi-vessel CAD (≥ 2 vessels >70% stenosis) and history of angina
* Chronic Obstructive Pulmonary Disease (COPD) with FEV1<50
* Permanent contralateral cranial nerve injury/paralysis
* Restenosis from previous carotid endarterectomy (CEA)
* Planned coronary artery bypass grafting (CABG) or valve replacement surgery between 31-60 days after CAS
* Abdominal aortic aneurysm surgical repair or Endovascular repair is planned between 31 to 60 days after CAS.

Anatomic conditions:

* Occlusion of the contralateral CCA or ICA.
* Prior radiation treatment to the neck or a radical neck dissection.
* Severe bilateral ICA stenosis requiring treatment.
* Target lesion at or above the level of the jaw (C2) or below the clavicle.
* Severe tandem lesions
* Inability to extend the neck due to cervical disorders.
* Laryngeal palsy or laryngectomy.
* Prior head and neck surgery in the region of the carotid artery.
* Tracheostomy or tracheostoma.
* Spinal immobility of the neck.
* Hostile neck or surgically inaccessible lesion.
* Target vessel and lesion meet all requirements for the CGuard Prime™ 80 stent:
* Target lesion location at the carotid bifurcation and/or proximal internal carotid artery (ICA)
* The diameter at the stent landing zone is between 4.8 mm and 9.0 mm.
* The target lesion length is ≤ 36 mm and can be covered by a single CGuard Prime™ 80 stent.
* Patient must have a 5 cm long disease-free segment of the common carotid artery (CCA) measured from the clavicle to the carotid bifurcation, with a minimum vessel diameter of 6 mm suitable for vascular access, sheath insertion, and vessel clamping.

EXCLUSION CRITERIA: Patients are not eligible for the study if they have any of the following exclusion criteria.

* Patient had or will have an interventional procedure or surgery of the carotid, coronary or peripheral arteries within 30 days before or after the index carotid procedure.
* Patient had or will have open heart surgery or valvular intervention (percutaneous or surgical), or any major operation, within 30 days before or after the index carotid procedure.
* Vascular anatomy that would preclude safe sheath insertion or deliverability of stent
* Patient had a previously placed stent in the ipsilateral ICA or CCA.
* Total occlusion or presence of a "string sign" of the ipsilateral ICA or CCA.
* Presence of a filling defect of the target lesion.
* Tandem lesions, which cannot be covered by a single CGuard Prime™ stent.
* Patient has a stenosis of the innominate artery or proximal CCA requiring revascularization
* Patient has an open neck stoma.
* Patient has a history of bleeding diatheses or coagulopathy.
* Patient has hypercoagulable state.
* Patient has an alternative source of cerebral embolus, including but not limited to:

  1. Chronic atrial fibrillation.
  2. Episode(s) of paroxysmal atrial fibrillation within the past 6 months or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
  3. Knowledge of cardiac sources of embolus (e.g. left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma).
  4. Recently (<60 days) implanted heart valve (either surgically or endovascularly) as a known source of emboli as confirmed on echocardiogram,
  5. Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis (as determined by angiography or CTA/MRA 6 months prior to index procedure) greater in severity than the lesion to be treated; cerebral aneurysm > 5mm; AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
* Patient has a known sensitivity or allergy to nickel or titanium.
* Patient has a sensitivity to contrast media that cannot be adequately pre-treated.
* Patient has a sensitivity to both forms of protocol-acceptable anticoagulation strategies (i.e., both heparin AND Bivalirudin)
* Patient has a sensitivity to an antiplatelet agent AND all protocol acceptable alternative antiplatelet options
* Patient has a known intolerance to statins.
* Patient has a life expectancy of less than 3 years from the date of enrollment as determined by the Wallaert Life Expectancy Scale
* Patient has malignancy, primary or recurrent, and does not have independent assessment of life expectancy performed by the treating oncologist or an appropriate specialist other than the physician performing TCAR.
* Patient has an evolving stroke or intracranial hemorrhage, or a history of previous intracranial hemorrhage or brain surgery within the past 12 months.
* Patient had a recent stroke (≤ 7 days) placing him/her at risk of a hemorrhagic conversion during the index procedure.
* Patient has a history of a major stroke with a neurologic deficit (NIHSS of ≥ 15 or mRS ≥3).
* Patient had a TIA or amaurosis fugax or stroke within 48 hours of the index procedure.
* Female patient who is pregnant or lactating or is planning to become pregnant.
* Dementia or other neurologic condition that is likely to confound the neurologic assessment.
* Clinical condition that, in the opinion of the investigator, makes endovascular therapy impossible or hazardous.
* Patient has been previously enrolled in this clinical trial.
* Patient is likely to be non-compliant with protocol-required follow up or medication in the opinion of the investigator.
* Patient is currently participating in another clinical trial that has not completed its primary endpoint assessment or that may confound this study results.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Acute device success | From enrollment to end of follow-up at 1 year
  Successful insertion of the delivery system, successful deployment of the CGuard Prime™ 80 stent, and successful retraction of the delivery system when used in conjunction with the FDA-cleared ENROUTE NPS during a TCAR procedure.
Technical success | From enrollment to end of follow-up at 1 year
  Technical Success Rate is defined as the number of patients with at least one CGuard Prime™ 80 device successfully delivered and deployed with final residual diameter stenosis < 30% following final post-balloon dilatation (if performed) divided by the total number of patients where CGuard Prime™ 80 device deployment was attempted when used in conjunction with the FDA-cleared ENROUTE NPS during a TCAR procedure.

SECONDARY OUTCOMES:
Procedural success | From enrollment to 30-day follow-up
  Acute device success for CGuard PrimeTM 80 Delivery System and Stent without experiencing death, stroke or MI through 30-day post-procedure when used in conjunction with the FDA-cleared ENROUTE NPS during a TCAR procedure.
Treatment success | From enrollment to 30-day follow-up
  Treatment Success Rate is defined as the number of patients who meet CGuard Prime™ 80 Technical Success Rate without experiencing death, stroke or MI through 30-day post-procedure, divided by the total number of patients where CGuard Prime™ 80 device deployment was attempted when used in conjunction with the FDA-cleared ENROUTE NPS during a TCAR procedure.
Occurence of Hierarchical Death, Stroke or Myocardial Infarction (DSMI) within 30 days of the procedure | From enrollment to 30-day follow-up
Hierarchical Death or Stroke rate within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of death within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of all strokes within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of major stroke within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of minor stroke within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of Myocardial Infarction (MI) within 30 days of the procedure | From enrollment to 30-day follow-up
Rate of stent thrombosis or occlusion within 30 days of the index procedure | From enrollment to 30-day follow-up
Rate of stent thrombosis or occlusion through 1-year of the index procedure | From enrollment to end of follow-up at 1 year
All device-related serious adverse events within 30 days of the procedure | From enrollment to 30-day follow-up
All device-related serious adverse events through 1-year of the procedure | From enrollment to end of follow-up at 1 year
Rate of ipsilateral strokes between 31- and 365-day post index procedure | From time of 30-day follow-up to end of follow-up at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Geraghty, MD, Principal Investigator — Washington University School of Medicine; Patrick E. Muck, MD, Principal Investigator — TriHealth Inc.
Locations (8):
- United States (8):
  - UC Davis Health, Sacramento, California
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Allina, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Benefis Health System, Great Falls, Montana
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - TriHealth, Cincinnati, Ohio